CLINICAL TRIAL: NCT02105701
Title: A Phase III Randomized Clinical Trial to Study the Efficacy and Safety of the Combination Regimen of MK-5172/MK-8742 in Subjects Who Have Failed Prior Treatment With Pegylated Interferon and Ribavirin (P/R) With Chronic HCV GT1, GT4, and GT6 Infection
Brief Title: Study of Efficacy and Safety of Grazoprevir (MK-5172) + Elbasvir (MK-8742) With or Without Ribavirin for Participants With Hepatitis C Genotype 1, 4, or 6 Infections Who Have Failed Prior Treatment With Pegylated Interferon + Ribavirin (MK-5172-068)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5172-068; 2014-000824-12 (EudraCT Number)
Record Dates: First submitted 2014-04-02; First posted 2014-04-07 (Estimated); Results first posted 2016-03-04 (Estimated); Last update posted 2021-02-05 (Actual); Status verified 2021-01

CONDITIONS: Hepatitis C Infection
MeSH Terms: conditions — Hepatitis C | interventions — elbasvir-grazoprevir drug combination; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Grazoprevir + Elbasvir 12 weeks (Experimental): Participants receive grazoprevir 100 mg/elbasvir 50 mg fixed-dose combination (FDC) tablets once daily (q.d.) by mouth for 12 weeks.
  Interventions: Drug: Grazoprevir + Elbasvir
- Grazoprevir + Elbasvir + RBV 12 weeks (Experimental): Participants receive grazoprevir 100 mg/elbasvir 50 mg FDC tablets q.d. by mouth, along with RBV capsules twice daily (b.i.d.) by mouth (weight-based dosing; 800 to 1400 mg total daily dose), for 12 weeks.
  Interventions: Drug: Grazoprevir + Elbasvir; Drug: Ribavirin
- Grazoprevir + Elbasvir 16 weeks (Experimental): Participants receive grazoprevir 100 mg/elbasvir 50 mg FDC tablets q.d. by mouth for 16 weeks.
  Interventions: Drug: Grazoprevir + Elbasvir
- Grazoprevir + Elbasvir + RBV 16 weeks (Experimental): Participants receive grazoprevir 100 mg/elbasvir 50 mg FDC tablets q.d. by mouth, along with RBV capsules b.i.d. by mouth (weight-based dosing; 800 to 1400 mg total daily dose), for 16 weeks.
  Interventions: Drug: Grazoprevir + Elbasvir; Drug: Ribavirin

INTERVENTIONS:
Drug: Grazoprevir + Elbasvir — FDC tablet containing grazoprevir 100 mg and elbasvir 50 mg.
  Other Names: MK-5172A
Drug: Ribavirin — 200 mg capsule
  Other Names: Rebetol®
  Arms: Grazoprevir + Elbasvir + RBV 12 weeks; Grazoprevir + Elbasvir + RBV 16 weeks

SUMMARY:
This is an efficacy and safety study of grazoprevir (MK-5172) in combination with elbasvir (MK-8742) with or without ribavirin (RBV) in participants with chronic hepatitis C virus (HCV) genotype (GT) 1, 4, or 6 infections who have failed prior therapy with pegylated interferon and RBV. The primary study hypothesis is that in at least one of the study arms, the percentage of participants achieving sustained viral response 12 weeks after the end of all study treatment (SVR12) will be superior to 58%.

ELIGIBILITY:
Inclusion Criteria:

* Documented chronic HCV GT1, GT4, or GT6 with no evidence of non-typable or mixed genotype infection (positive for anti-HCV antibody, HCV ribonucleic acid [RNA], or any of the listed GTs at least 6 months prior to screening must be confirmed by screening lab results)
* Cirrhosis defined as liver biopsy showing METAVIR F4; or Fibroscan showing result >12.5 kilopascals (kPa); or FibroSure® (Fibrotest®) score of >0.75 and an aspartate aminotransferase (AST):platelet ratio index (APRI) of >2
* Absence of cirrhosis defined as liver biopsy showing absence of cirrhosis; or Fibroscan result of ≤ 12.5 kPa; or Fibrosure® (Fibrotest®) score of ≤ 0.48 and APRI ≤ 1
* Previous HCV treatment status of peginterferon/RBV Null responder; or peginterferon/RBV Partial responder; or peginterferon/RBV Treatment Relapse
* For human immunodeficiency virus (HIV) co-infected participants: documented HIV-1 infection; currently naïve to treatment with any antiretroviral therapy (ART) and have no plans to initiate ART treatment while participating in this study; or be on HIV ART for at least 8 weeks prior to study entry (dual nucleoside reverse transcriptase inhibitor [NRTI] backbone of tenofovir or abacavir and either emtricitabine or lamivudine plus raltegravir (or dolutegravir or rilpivirine) (no changes in HIV regimen allowed within 4 weeks of randomization); cluster of differentiation 4 (CD4)+ T-cell count >200 cells/mm^3 at screening; documented undetectable plasma HIV-1 RNA at least 8 weeks prior to screening; participants not on ART, HIV RNA must be <50,000 copies/mL; must have at least one viable antiretroviral regimen alternative beyond their current regimen in the event of HIV virologic failure and the development of antiretroviral drug resistance
* Agree to use two acceptable methods of birth control from at least 2 weeks prior to Day 1 and continue until at least 6 months after last dose of study drug, or longer if dictated by local regulations; a male participant who is not (or whose partner is not) of reproductive potential is eligible without requiring the use of contraception

Exclusion Criteria:

* Evidence of decompensated liver disease manifested by the presence of or history of ascites, esophageal or gastric variceal bleeding, hepatic encephalopathy or other signs or symptoms of advanced liver disease
* For participants with cirrhosis, participants who are Child-Pugh Class B or C or who have a Pugh-Turcotte (CPT) score >6, must be excluded
* Co-infected with hepatitis B virus
* Has had previous direct-acting antiviral treatment
* History of malignancy <=5 years prior except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer or carcinoma in situ; or is under evaluation for other active or suspected malignancy
* Has cirrhosis and liver imaging showing evidence of hepatocellular carcinoma (HCC) or is under evaluation for HCC
* Taking or plans to take any HIV therapy that includes a ritonavir-boosted or unboosted protease inhibitor, efavirenz or etravirine
* Currently participating or has participated in a study with an investigational compound within 30 days of signing informed consent and is not willing to refrain from participating in another such study during the course of this study
* Clinically-relevant drug or alcohol abuse within 12 months
* Pregnant, breast-feeding, or expecting to conceive or donate eggs or sperm from Day 1 and continue until at least 6 months after last dose of study drug, or longer if dictated by local regulations; or is a male whose female partner(s) is/are pregnant
* History of organ transplant (including hematopoietic stem cell transplants) other than cornea and hair
* Poor venous access
* History of gastric surgery (e.g., stapling, bypass) or history of malabsorption disorders (e.g., celiac sprue disease)
* Hemoglobinopathy, including, but not limited to, thalassemia major
* Any medical condition requiring, or likely to require, chronic systemic corticosteroids, tumor necrosis factor (TNF) antagonists, or other immunosuppressant drugs during the course of the trial
* For participants with HIV, history of opportunistic infection in the preceding 6 months
* For participants with HIV, use of HIV drugs other than a dual NRTI backbone of tenofovir or abacavir and either emtricitabine or lamivudine plus raltegravir (or dolutegravir or rilpivirine)
* Evidence or history of chronic hepatitis not caused by HCV, including but not limited to nonalcoholic steatohepatitis (NASH), drug-induced hepatitis, and autoimmune hepatitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2014-06-05 (Actual); Primary Completion 2015-03-24 (Actual); Study Completion 2015-06-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Kwo P, Gane EJ, Peng CY, Pearlman B, Vierling JM, Serfaty L, Buti M, Shafran S, Stryszak P, Lin L, Gress J, Black S, Dutko FJ, Robertson M, Wahl J, Lupinacci L, Barr E, Haber B. Effectiveness of Elbasvir and Grazoprevir Combination, With or Without Ribavirin, for Treatment-Experienced Patients With Chronic Hepatitis C Infection. Gastroenterology. 2017 Jan;152(1):164-175.e4. doi: 10.1053/j.gastro.2016.09.045. Epub 2016 Oct 5. PMID 27720838
- [Derived] Asselah T, Reesink H, Gerstoft J, de Ledinghen V, Pockros PJ, Robertson M, Hwang P, Asante-Appiah E, Wahl J, Nguyen BY, Barr E, Talwani R, Serfaty L. Efficacy of elbasvir and grazoprevir in participants with hepatitis C virus genotype 4 infection: A pooled analysis. Liver Int. 2018 Sep;38(9):1583-1591. doi: 10.1111/liv.13727. Epub 2018 Mar 31. PMID 29461687
- [Derived] Reau N, Robertson MN, Feng HP, Caro L, Yeh WW, Nguyen BT, Wahl J, Barr E, Hwang P, Klopfer SO. Concomitant proton pump inhibitor use does not reduce the efficacy of elbasvir/grazoprevir: A pooled analysis of 1,322 patients with hepatitis C infection. Hepatol Commun. 2017 Aug 22;1(8):757-764. doi: 10.1002/hep4.1081. eCollection 2017 Oct. PMID 29404492
- [Derived] Jacobson IM, Lawitz E, Kwo PY, Hezode C, Peng CY, Howe AYM, Hwang P, Wahl J, Robertson M, Barr E, Haber BA. Safety and Efficacy of Elbasvir/Grazoprevir in Patients With Hepatitis C Virus Infection and Compensated Cirrhosis: An Integrated Analysis. Gastroenterology. 2017 May;152(6):1372-1382.e2. doi: 10.1053/j.gastro.2017.01.050. Epub 2017 Feb 11. PMID 28193518

RESULTS

PARTICIPANT FLOW:
Groups:
- Grazoprevir + Elbasvir 12 Weeks: Participants received grazoprevir 100 mg/elbasvir 50 mg FDC tablets q.d. by mouth for 12 weeks.
- Grazoprevir + Elbasvir + RBV 12 Weeks: Participants received grazoprevir 100 mg/elbasvir 50 mg FDC tablets q.d. by mouth, along with RBV capsules b.i.d. by mouth (weight-based dosing; 800 to 1400 mg total daily dose), for 12 weeks.
- Grazoprevir + Elbasvir 16 Weeks: Participants received grazoprevir 100 mg/elbasvir 50 mg FDC tablets q.d. by mouth for 16 weeks.
- Grazoprevir + Elbasvir + RBV 16 Weeks: Participants received grazoprevir 100 mg/elbasvir 50 mg FDC tablets q.d. by mouth, along with RBV capsules b.i.d. by mouth (weight-based dosing; 800 to 1400 mg total daily dose), for 16 weeks.
Period: Overall Study
Arm/Group | Grazoprevir + Elbasvir 12 Weeks | Grazoprevir + Elbasvir + RBV 12 Weeks | Grazoprevir + Elbasvir 16 Weeks | Grazoprevir + Elbasvir + RBV 16 Weeks
Started | 105 | 104 | 105 | 106
Completed | 101 | 103 | 102 | 104
Not Completed | 4 | 1 | 3 | 2
Not completed — Lost to Follow-up | 1 | 0 | 2 | 1
Not completed — Protocol Violation | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 0 | 1
Not completed — Death | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Grazoprevir + Elbasvir 12 Weeks | Grazoprevir + Elbasvir + RBV 12 Weeks | Grazoprevir + Elbasvir 16 Weeks | Grazoprevir + Elbasvir + RBV 16 Weeks | Total
Number analyzed (Participants) | 105 | 104 | 105 | 106 | 420
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.71 (9.81) | 55.46 (8.26) | 54.91 (9.79) | 54.98 (9.61) | 55.27 (9.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 32 | 36 | 42 | 149
  Male | 66 | 72 | 69 | 64 | 271

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Undetectable HCV RNA 12 Weeks After Completing Study Therapy (SVR12)
Description: HCV RNA was measured using the Roche COBAS® Taqman® HCV Test, v2.0 assay.
Time Frame: 12 weeks after the end of all study treatment (up to 28 weeks)
Population: The Full Analysis Set (FAS) population consists of all randomized subjects who receive at least one dose of study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Grazoprevir + Elbasvir 12 Weeks | Grazoprevir + Elbasvir + RBV 12 Weeks | Grazoprevir + Elbasvir 16 Weeks | Grazoprevir + Elbasvir + RBV 16 Weeks
Number analyzed (Participants) | 105 | 104 | 105 | 106
Percentage of participants | 92.4 [85.5 to 96.7] | 94.2 [87.9 to 97.9] | 92.4 [85.5 to 96.7] | 98.1 [93.4 to 99.8]
Statistical Analysis 1: Comparison: Grazoprevir + Elbasvir 12 Weeks; The hypothesis was that at least 1 treatment arm would have a SVR12 rate >58%; Test type: Superiority or Other; p < 0.001, One-sided Exact Test
Statistical Analysis 2: Comparison: Grazoprevir + Elbasvir + RBV 12 Weeks; The hypothesis was that at least 1 treatment arm would have a SVR12 rate >58%; Test type: Superiority or Other; p < 0.001, One-sided Exact Test
Statistical Analysis 3: Comparison: Grazoprevir + Elbasvir 16 Weeks; The hypothesis was that at least 1 treatment arm would have a SVR12 rate >58%; Test type: Superiority or Other; p < 0.001, One-sided Exact Test
Statistical Analysis 4: Comparison: Grazoprevir + Elbasvir + RBV 16 Weeks; The hypothesis was that at least 1 treatment arm would have a SVR12 rate >58%; Test type: Superiority or Other; p < 0.001, One-sided Exact Test

2. Primary Outcome: Number of Participants Experiencing Adverse Events (AE)
Description: An AE is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment.
Time Frame: Up to 18 weeks
Population: The All Participants as Treated (APaT) population consists of all participants who received at least one dose of study treatment.
Measure: Number; unit: Number of participants
Arm/Group | Grazoprevir + Elbasvir 12 Weeks | Grazoprevir + Elbasvir + RBV 12 Weeks | Grazoprevir + Elbasvir 16 Weeks | Grazoprevir + Elbasvir + RBV 16 Weeks
Number analyzed (Participants) | 105 | 104 | 105 | 106
Number of participants | 74 | 85 | 77 | 95

3. Primary Outcome: Number of Participants Discontinuing Study Treatment Due to an AE
Description: as for outcome 2
Time Frame: Up to 16 weeks
Population: as for outcome 2
Measure: Number; unit: Number of participants
Arm/Group | Grazoprevir + Elbasvir 12 Weeks | Grazoprevir + Elbasvir + RBV 12 Weeks | Grazoprevir + Elbasvir 16 Weeks | Grazoprevir + Elbasvir + RBV 16 Weeks
Number analyzed (Participants) | 105 | 104 | 105 | 106
Number of participants | 1 | 1 | 0 | 5

4. Secondary Outcome: Percentage of Participants Achieving Undetectable HCV RNA 24 Weeks After the End of All Treatment (SVR24)
Description: HCV RNA was measured using the Roche COBAS® Taqman® HCV Test, v2.0 assay.
Time Frame: 24 weeks after the end of all study treatment (up to 40 weeks)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Grazoprevir + Elbasvir 12 Weeks | Grazoprevir + Elbasvir + RBV 12 Weeks | Grazoprevir + Elbasvir 16 Weeks | Grazoprevir + Elbasvir + RBV 16 Weeks
Number analyzed (Participants) | 105 | 104 | 105 | 106
Percentage of participants | 91.4 [84.4 to 96.0] | 94.2 [87.9 to 97.9] | 89.5 [82.0 to 94.7] | 95.3 [89.3 to 98.5]
Statistical Analysis 1: Comparison: Grazoprevir + Elbasvir 12 Weeks; The hypothesis was that at least 1 treatment arm would have a SVR24 rate >58%; Test type: Superiority or Other; p < 0.001, One-sided Exact Test
Statistical Analysis 2: Comparison: Grazoprevir + Elbasvir + RBV 12 Weeks; The hypothesis was that at least 1 treatment arm would have a SVR24 rate >58%; Test type: Superiority or Other; p < 0.001, One-sided Exact Test
Statistical Analysis 3: Comparison: Grazoprevir + Elbasvir 16 Weeks; The hypothesis was that at least 1 treatment arm would have a SVR24 rate >58%; Test type: Superiority or Other; p < 0.001, One-sided Exact Test
Statistical Analysis 4: Comparison: Grazoprevir + Elbasvir + RBV 16 Weeks; The hypothesis was that at least 1 treatment arm would have a SVR24 rate >58%; Test type: Superiority or Other; p < 0.001, One-sided Exact Test

ADVERSE EVENTS:
Time Frame: Up to Week 40.
Description: An AE is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment.
Groups:
- GZR/EBR 12 Weeks: Participants received grazoprevir 100 mg/elbasvir 50 mg FDC tablets q.d. by mouth for 12 weeks.
- GZR/EBR + RBV 12 Weeks: Participants received grazoprevir 100 mg/elbasvir 50 mg FDC tablets q.d. by mouth, along with RBV capsules b.i.d. by mouth (weight-based dosing; 800 to 1400 mg total daily dose), for 12 weeks.
- GZR/EBR 16 Weeks: Participants received grazoprevir 100 mg/elbasvir 50 mg FDC tablets q.d. by mouth for 16 weeks.
- GZR/EBR + RBV for 16 Weeks: Participants received grazoprevir 100 mg/elbasvir 50 mg FDC tablets q.d. by mouth, along with RBV capsules b.i.d. by mouth (weight-based dosing; 800 to 1400 mg total daily dose), for 16 weeks.
Arm/Group | GZR/EBR 12 Weeks | GZR/EBR + RBV 12 Weeks | GZR/EBR 16 Weeks | GZR/EBR + RBV for 16 Weeks
Serious Adverse Events (participants affected / at risk) | 6/105 | 8/104 | 4/105 | 6/106
Other Adverse Events (participants affected / at risk) | 55/105 | 72/104 | 58/105 | 84/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GZR/EBR 12 Weeks (N=105) | GZR/EBR + RBV 12 Weeks (N=104) | GZR/EBR 16 Weeks (N=105) | GZR/EBR + RBV for 16 Weeks (N=106)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sudden hearing loss (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal angioedema (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Varices oesophageal (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes simplex oesophagitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infectious colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Parotitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Splenic marginal zone lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Schizophrenia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Uterine polyp (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Femoral artery occlusion (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GZR/EBR 12 Weeks (N=105) | GZR/EBR + RBV 12 Weeks (N=104) | GZR/EBR 16 Weeks (N=105) | GZR/EBR + RBV for 16 Weeks (N=106)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 12 (13) | 0 (0) | 17 (19)
Abdominal pain (Gastrointestinal disorders) | 6 (6) | 3 (3) | 1 (1) | 3 (3)
Constipation (Gastrointestinal disorders) | 1 (1) | 3 (3) | 7 (8) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 4 (4) | 8 (9) | 9 (9)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 4 (4) | 0 (0) | 7 (9)
Nausea (Gastrointestinal disorders) | 9 (10) | 15 (19) | 4 (4) | 18 (20)
Vomiting (Gastrointestinal disorders) | 2 (2) | 7 (8) | 1 (1) | 9 (10)
Asthenia (General disorders) | 8 (9) | 11 (13) | 9 (10) | 10 (10)
Fatigue (General disorders) | 20 (21) | 28 (32) | 17 (18) | 32 (33)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 2 (2) | 6 (9) | 5 (6)
Accidental overdose (Injury, poisoning and procedural complications) | 3 (3) | 15 (22) | 1 (1) | 14 (23)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 7 (7)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 6 (6) | 1 (1) | 6 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (4) | 7 (8) | 4 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 6 (7) | 8 (8) | 7 (7)
Dizziness (Nervous system disorders) | 7 (7) | 8 (8) | 5 (10) | 6 (8)
Headache (Nervous system disorders) | 21 (23) | 21 (23) | 21 (23) | 20 (22)
Insomnia (Psychiatric disorders) | 5 (5) | 11 (12) | 7 (7) | 10 (10)
Irritability (Psychiatric disorders) | 4 (6) | 5 (5) | 2 (2) | 8 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 10 (10) | 4 (4) | 10 (10)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 9 (11) | 1 (1) | 10 (10)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (4) | 0 (0) | 8 (8)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 11 (13) | 6 (6) | 11 (11)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 4 (4) | 1 (1) | 8 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation.